CLINICAL TRIAL: NCT03421236
Title: Intravesical Ty21a for the Treatment of Patients With Non-muscle-invasive Bladder Cancer (NMIBC)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Patrice Jichlinski (Other)
Responsible Party: Sponsor-Investigator, Patrice Jichlinski, Professor, Dpt Chief, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IvesTy21a
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Non Muscle Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Ty21a typhoid vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- non muscle invasive bladder cancer patient (Experimental): intravesical instillation of Ty21a in patients not requiring BCG
  Interventions: Biological: Ty21a

INTERVENTIONS:
Biological: Ty21a — intravesical administration of Ty21a

SUMMARY:
Bladder cancer is the fourth and eighth most common malignancy among men and women, respectively. About 75% of bladder cancers are diagnosed as non muscle-invasive and according to specific tumor-stage and grade characteristics, intravesical immunotherapy with Bacillus Calmette-Guérin (BCG) is used to prevent recurrence and/or progression. However, BCG immunotherapy is associated with significant adverse events and treatment failure may occur in 30-40% of cases, hence the necessity for alternative therapies. In an orthotopic MB49 mouse bladder cancer model, another bacterial vaccine (Ty21a/Vivotif) turned out to be more effective than BCG for inducing tumor regression and mice survival upon intravesical instillation; and potentially safer because Ty21a bacteria did not infect/persist in any mice tissues nor in human bladder explants or cell lines, in contrast to BCG. Ty21a/Vivotif has been used in the last 30 years in millions of individuals as an oral typhoid vaccine with a high safety record. In this phase I trial we will be testing the safety of intravesical administration of Ty21a and its effect on bladder immunity in non-muscle invasive bladder cancer (NMIBC) patients, for whom recommendation of BCG therapy is not mandatory.

DETAILED DESCRIPTION:
Escalating doses of Ty21a/Vivotif® will be administered by the intravesical route to evaluate whether Ty21 may replace the standard BCG immunotherapy in NMIBC patients.

The minimal starting dose will be instilled intravesically once a week for 4 weeks in 3 patients. If well tolerated, a 5-fold higher dose will be instilled 4-times in 3 other patients, and so on for a maximum of 4 doses to be tested.

The maximal tolerated dose will then be administered to 3 new patients 6-times once a week. If 6 instillations are well tolerated, 7 additional patients will be included to receive 6 instillations with this maximal tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an intermediary or low risk of progression of bladder cancer (according to an EORTC score and clinical considerations) and thus not requiring BCG immunotherapy will be included after a transurethral resection of the bladder tumor (TURBT). Male and Female patients aged > 18yrs, with a Karnofsky performance status of 60% or more, sero-negative for HIV, HBV and HCV and with laboratory parameters for vital function in the normal range or with abnormalities without clinical significance may be included.

Exclusion Criteria:

* Patients with NMIBC that require BCG treatments or with muscle-invasive bladder cancer, sero-positive for HIV, HBV and HCV or with other serious illnesses (e.g., serious infections requiring antibiotics, bleeding disorders, autoimmune disease), will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-02-18 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 6 weeks
  safety and tolerability of intravesical Ty21a

CONTACTS AND LOCATIONS:
Locations (1):
- Dpt Urology- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lucca I, Derre L, Cesson V, Bohner P, Crettenand F, Rodrigues-Dias S, Dartiguenave F, Masnada A, Texeira-Pereira C, Benmerzoug S, Chevalier M, Domingos-Pereira S, Nguyen S, Polak L, Schneider A, Roth B, Jichlinski P, Nardelli-Haefliger D. Intravesical Ty21a Treatment of Non-muscle-invasive Bladder Cancer Shows a Good Safety Profile. Eur Urol Open Sci. 2022 Oct 3;45:55-58. doi: 10.1016/j.euros.2022.09.004. eCollection 2022 Nov. PMID 36212980